CLINICAL TRIAL: NCT05204914
Title: Effect Of Supraglottic Airway Devices On The Tempromandibular Joint Function Following Prolonged General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya mohammed el_otafey, Principal investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Soh-med-21-10-05
Record Dates: First submitted 2021-12-09; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Change of Tempromandibular Joint Function With Supra Glottic Airway Devices
Keywords: The interincisors distance& movements of the jaw

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supra glottic airway devices (Other)
  Interventions: Device: Supra glottic airway devices

INTERVENTIONS:
Device: Supra glottic airway devices — Using the device in save air way in patients under general anesthesia and the change in the tempromandibular joint will be evaluated

SUMMARY:
Effect Of Supraglottic Airway Devices On The Tempromandibular Joint function Following Prolonged General Anesthesia

DETAILED DESCRIPTION:
Supraglottic airway devices (SADs) are used for securing the airway in over 50% of general anesthetics; They are used for both spontaneously & ventilated patients; They also used as conduits to aid endotracheal intubation when both positive mechanical ventilation ( PMV) & tradional endotracheal intubation( ETT) have failed

All (SADs) consist of a tube that connected to a breathing circuit or a breathing bag which is attached to a hypopharengeal device that seals air flow to the glottis

There are many types of SADs including I-Gel, intubating laryngeal mask airway (LMA), LMA CTrash and LMA proseal Although considered relatively safe devices; and have many advantages as they are less invasive than EET, less incidence of bronchospasm, don't often require muscle relaxation or neck mobility

There are several potential complications & disadvantages ; Include temporomandibular joint (TMJ) dysfunction, increases the risk of aspiration, more gas leak &pollution, less safe in prone postion & deeper anaethesia is required

This study will investigate (TMJ) dysfunction following the use of a (SAD) during general anesthesia, as There are a number of insertion maneuvers described for (SADs) [2] such as a jaw thrust may result in temporomandibular joint (TMJ) dysfunction by anteriorly displacing the mandible . In addition, other factors such as degree of muscle relaxation leading to hypotonicity of jaw muscles and passive mouth opening. In addition, for the duration of the operation the mouth is kept slightly open by a breathing tube may result in (TMJ) dislocation.

The inter-incisor distance will be measured using a Therabite â ruler (ATOS Medical, Nottingham, UK). This has a scale from 0 to 70 mm with 1-mm markings. The accuracy of this type of ruler is1.0 mm. The Therabite ruler was chosen as it routinely used by the investigators for (TMJ) assessment in the maxillofacial clinic.

ELIGIBILITY:
Inclusion The study will include 60 adult patients (>18 years old) with ASA physical status class I and class II scheduled for elective surgery under general anesthesia where SADs ara planned to be used as airway devices

Exclusion Criteria:

1. Patient refusal
2. limited mouth opening(<2 fingers)
3. Facial &upper airway trauma
4. Patients with dentures or who were edentulous (as accurate objective measurements would be difficult to determine)
5. Head and neck surgery (as surgery may influence TMJ function)
6. GITsurgery (as SAD doesn't completely protect air way against aspiration )
7. Pt with preexisting tempromadibular joint dysfunction
8. Duration of anaethesia less than 1 h or more than 4hs-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-30 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in tempromandibular jiont function | Single measurement Within 24 hours postoperative
  The change in inter incisors distance,forword movement&lat movement of the jow post operative will be measured also any post op pain or difficulty in movement of the jow will be recorded

SECONDARY OUTCOMES:
Other complications of supraglottic airway devices | Intra operative &24hours postoperative
  Including aspiration and airway edema